CLINICAL TRIAL: NCT05061719
Title: An Open-label, Multicenter Trial to Assess the Safety and Tolerability of Lumateperone as Adjunctive Therapy in the Treatment of Patients With Major Depressive Disorder
Brief Title: An Open-label Study of Lumateperone as Adjunctive Therapy in the Treatment of Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITI-007-503
Record Dates: First submitted 2021-09-20; First posted 2021-09-29 (Actual); Results first posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Major Depressive Disorder
Keywords: Adjunctive MDD Therapy
MeSH Terms: conditions — Depressive Disorder, Major | interventions — lumateperone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lumateperone 42 mg (Experimental)
  Interventions: Drug: Lumateperone

INTERVENTIONS:
Drug: Lumateperone — Lumateperone 42 mg capsules administered orally, once daily

SUMMARY:
This is a multicenter, open-label, fixed dose, 26 week study of patients with MDD. Eligible patients from the lead-in studies will enter the Open-label Safety Study at the Screening/Baseline Visit (Visit 1/Day 1), at which point patient eligibility will be assessed and informed consent obtained.

DETAILED DESCRIPTION:
At the Screening/Baseline Visit (Visit 1/Day 1), which is the same visit as Visit 8/Day 43 of the lead-in study, eligible patients will receive open-label lumateperone 42 mg once daily for approximately 26 weeks. Patients will continue their background ADT from the lead-in study. Patients will be seen for weekly visits through Visit 5/Week 4. Thereafter, visits will occur every two weeks. A Safety Follow-up visit will occur on Visit 17/Day 197, approximately 2 weeks after the last dose of open-label lumateperone 42 mg.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the Investigator, patients must have safely completed the lead-in study.
2. Patient is taking their ADT as prescribed from the lead-in study.

Exclusion Criteria:

1. In the opinion of the Investigator, the patient is unable to comply with study procedures or judged to be inappropriate for the study.
2. In the opinion of the Investigator, the patient has a significant risk for suicidal behavior during the course of her/his participation in the study or is considered to be an imminent danger to her/himself or others, and/or:

   1. At the Screening/Baseline Visit, the patient scores "yes" on Suicidal Ideation Items 4 or 5 of the C SSRS "Since Last Visit" version;
   2. At the Screening/Baseline visit, the patient scores ≥ 5 on the MADRS Item 10 (Suicidal Thoughts).
3. Based on the Investigator's clinical judgement, any abnormal clinical laboratory test or ECG results obtained throughout the lead-in study that are considered clinically significant and preclude safe participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 812 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-10-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (96):
- United States (38):
  - Clinical Site, Phoenix, Arizona
  - Clinical Site, Bentonville, Arkansas
  - Clinical Site, Little Rock, Arkansas
  - Clinical Site, Rogers, Arkansas
  - Clinical Site, Culver City, California
  - Clinical Site, Glendale, California
  - Clinical Site, Newport Beach, California
  - Clinical Site, Oceanside, California
  - Clinical Site, Redlands, California
  - Clinical Site, Riverside, California
  - Clinical Site, San Diego, California
  - Clinical Site, Sherman Oaks, California
  - Clinical Site, Temecula, California
  - Clinical Site, Upland, California
  - Clinical Site, Fort Lauderdale, Florida
  - Clinical Site, Jacksonville, Florida
  - Clinical Site, Orlando, Florida
  - Clinical Site, Palm Bay, Florida
  - Clinical Site, West Palm Beach, Florida
  - Clinical Site, Atlanta, Georgia
  - Clinical Site, Decatur, Georgia
  - Clinical Site, Joliet, Illinois
  - Clinical Site, Overland Park, Kansas
  - Clinical Site, Gaithersburg, Maryland
  - Clinical Site, Boston, Massachusetts
  - Clinical Site, Flowood, Mississippi
  - Clinical Site, Saint Charles, Missouri
  - Clinical Site, Berlin, New Jersey
  - Clinical Site, Toms River, New Jersey
  - Clinical Site, Brooklyn, New York
  - Clinical Site, Cedarhurst, New York
  - Clinical Site, Mount Kisco, New York
  - Clinical Site, Charlotte, North Carolina
  - Clinical Site, Allentown, Pennsylvania
  - Clinical Site, Media, Pennsylvania
  - Clinical Site, Plymouth Meeting, Pennsylvania
  - Clinical Site, Austin, Texas
  - Clinical Site, Bellevue, Washington
- Bulgaria (11):
  - Clinical Site, Burgas
  - Clinical Site, Kazanlak
  - Clinical Site, Novi Iskar
  - Clinical Site, Pleven
  - Clinical Site, Plovdiv
  - Clinical Site, Rousse
  - Clinical Site, Sofia
  - Clinical Site, Targovishte
  - Clinical Site, Tsarev Brod
  - Clinical Site, Veliko Tarnovo
  - Clinical Site, Vratsa
- Czechia (6):
  - Clinical Site, Brno
  - Clinical site, Brno
  - Clinical Site, Hostivice
  - Clinical Site, Ostrava
  - Clinical Site, Pilsen
  - Clinical Site, Prague
- Finland (2):
  - Clinical Site, Helsinki
  - Clinical Site, Oulu
- Germany (6):
  - Clinical Site, Bad Homburg
  - Clinical Site, Freiburg im Breisgau
  - Clinical Site, Hamburg
  - Clinical Site, Mittweida
  - Clinical Site, Schwerin
  - Clinical Site, Westerstede
- Hungary (3):
  - Clinical Site, Budapest
  - Clinical Site, Debrecen
  - Clinical Site, Gyöngyös
- India (10):
  - Clinical Site, Guwahati, Assam
  - Clinical Site, Ahmedabad, Gujarat
  - Clinical Site, Jūnāgadh, Gujarat
  - Clinical Site, Vadodara, Gujarat
  - Clinical Site, Mysore, Karnataka
  - Clinical Site, Aurangabad, Maharashtra
  - Clinical Site, Nagpur, Maharashtra
  - Clinical Site, Nashik, Maharashtra
  - Clinical Site, Mumbai
  - Clinical Site, Nashik
- Poland (9):
  - Clinical Site, Bełchatów
  - Clinical Site, Bialystok
  - Clinical Site, Bydgoszcz
  - Clinical Site, Gdansk
  - Clinical Site, Gorlice
  - Clinical Site, Leszno
  - Clinical Site, Pruszcz Gdański
  - Clinical SIte, Torun
  - Clinical Site, Wroclaw
- Slovakia (6):
  - Clinical Site, Bratislava
  - Clinical Site, Košice
  - Clinical Site, Rimavská Sobota
  - Clinical Site, Svidník
  - Clinical Site, Vranov nad Topľou
  - Clinical Site, Zlaté Moravce
- South Korea (3):
  - Clinical Site, Ansan-si, North Chungcheong
  - Clinical Site, Gwangju
  - Clinical Site, Seoul
- Sweden (2):
  - Clinical Site, Lund
  - Clinical Site, Stockholm

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 812 patients were enrolled; 809 patients received at least one dose of study drug and included in the Safety Population.
Period: Overall Study
Arm/Group | Lumateperone 42 mg
Started | 809
Completed | 684
Not Completed | 125
Not completed — Adverse Event | 60
Not completed — Death | 1
Not completed — Lack of Efficacy | 7
Not completed — Lost to Follow-up | 5
Not completed — Pregnancy | 1
Not completed — Protocol Violation | 8
Not completed — Withdrawal by Subject | 41
Not completed — Site Closure | 2

BASELINE CHARACTERISTICS:
Arm/Group | Lumateperone 42 mg
Number analyzed (Participants) | 809
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (12.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 549
  Male | 260
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 703
  Black or African American | 37
  Asian | 61
  Native Hawaiian or Other Pacific Islander | 2
  Multiple | 4
  Other | 2
Region of Enrollment [Number; unit: participants]
  Sweden | 2
  Hungary | 15
  United States | 225
  Czechia | 95
  Poland | 147
  Slovakia | 32
  Bulgaria | 159
  Germany | 25
  India | 53
  Argentina | 56

OUTCOME MEASURES:

1. Primary Outcome: The Number and Percentage of Patients Reporting Treatment Emergent Adverse Events
Description: An AE that occurs during the Open-label Treatment Period will be considered a treatment-emergent AE (TEAE) if it was not present before the date of the first dose of open-label lumateperone or was present before the date of the first dose of open-label lumateperone but changed in severity during the Open-label Treatment Period.
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lumateperone 42 mg
Number analyzed (Participants) | 809
Participants | 548

2. Secondary Outcome: Change From Baseline in One of the 6 Week Double-blind Lead-in Studies (NCT04985942 & NCT05061706) to the End of the Open-Label Treatment Period (a Combined Total of up to 32 Weeks) in the Montgomery-Åsberg Depression Rating Scale
Description: The MADRS is a clinician-rated 10 item scale to assess depressive symptoms. Each item is rated on a 7-point scale from 0-6. The total score ranges from 0 to 60 with a higher score indicating increased severity of depressive symptoms.
Time Frame: 32 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumateperone 42 mg
Number analyzed (Participants) | 809
score on a scale | -21.7 (8.39)

3. Secondary Outcome: Change From Baseline in One of the 6 Week Double-blind Lead-in Studies (NCT04985942 & NCT05061706) to the End of the Open-Label Treatment Period (a Combined Total of up to 32 Weeks) in the Clinical Global Impression Scale-Severity
Description: The CGI-S is a clinician-rated scale to assess a patient's overall mental health. The scale ranges from 1 (normal, not ta all ill) to 7 (among the most extremely ill patients).
Time Frame: 32 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumateperone 42 mg
Number analyzed (Participants) | 809
score on a scale | -2.5 (1.19)

ADVERSE EVENTS:
Time Frame: From signing ICF until end of study procedures (~28 weeks), including 26 weeks of open-label treatment.
Arm/Group | Lumateperone 42 mg
All-Cause Mortality (participants affected / at risk) | 1/809
Serious Adverse Events (participants affected / at risk) | 8/809
Other Adverse Events (participants affected / at risk) | 322/809
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lumateperone 42 mg (N=809)
Alcohol Poisoning (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2
Biliary colic (Hepatobiliary disorders) | 1
Helicobacter gastritis (Infections and infestations) | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lumateperone 42 mg (N=809)
Headache (Nervous system disorders) | 134
Dizziness (Nervous system disorders) | 86
Dry mouth (Gastrointestinal disorders) | 65
Nausea (Gastrointestinal disorders) | 62
Somnolence (Nervous system disorders) | 58
Diarrhoea (Gastrointestinal disorders) | 50
Nasopharyngitis (Infections and infestations) | 42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/19/NCT05061719/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-24): https://cdn.clinicaltrials.gov/large-docs/19/NCT05061719/SAP_001.pdf